CLINICAL TRIAL: NCT04927364
Title: Examining the Effectiveness of Deep TMS in Veterans With Alcohol Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Palo Alto Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Claudia Beatriz Padula, Health Research Science Specialist, VA Palo Alto Health Care System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 54988
Record Dates: First submitted 2021-06-01; First posted 2021-06-16 (Actual); Results first posted 2024-07-10 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Alcohol Use Disorder (AUD); Transcranial Magnetic Stimulation
Keywords: Veterans; Deep Transcranial Magnetic Stimulation (dTMS); Alcohol Use Disorder; Neuroimaging; Relapse
MeSH Terms: conditions — Alcoholism; Recurrence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Active dTMS (Experimental): Participants will receive 30 dTMS treatments, administered 3 times per day over 10 consecutive business days, Each treatment visit will last approximately 30 minutes in total.
  Interventions: Device: Deep Transcranial Magnetic Stimulation (dTMS) H7 coil

INTERVENTIONS:
Device: Deep Transcranial Magnetic Stimulation (dTMS) H7 coil — The study will utilize the H7 coil to administer Deep Transcranial Magnetic Stimulation (dTMS) to the dorsal anterior cingulate cortex (dACC), a core salience network node.

SUMMARY:
This study aims to evaluate the efficacy of deep transcranial magnetic stimulation (dTMS) as a treatment for Veterans with an alcohol use disorder (AUD).

DETAILED DESCRIPTION:
At least 60% of those with AUD will experience a major relapse period within 6 months of treatment, irrespective of the intervention (psychosocial and/or pharmacological) employed. Consequently, the high prevalence of AUD and relapse following treatment in Veterans is associated with substantial resource allocation and costs for the VA Health Care System. Current pharmacological and psychosocial interventions demonstrate only a moderate level of efficacy, which is reflected in the high rate of relapse in AUD.

TMS is a neurostimulation method that is at the forefront of innovative, non-invasive, and safe treatments for AUD, and other psychiatric disorders. To reduce the high rate of relapse in Veterans with AUD, it is necessary for interventions to more effectively address the associated neurobiological dysfunction. Non-invasive neuromodulation techniques are showing promise toward the aim of modifying specific and selective neural targets related to AUD and relapse. However, device-based interventions to date for AUD have focused on cortical stimulation. In contrast, preclinical and clinical studies, including our research team's preliminary data, suggest that subcortical nodes within the salience network could be promising novel neuromodulation targets. The dorsal anterior cingulate cortex (dACC) is a core node of the salience network, and hence the target of this proposal. Deep repetitive transcranial magnetic stimulation (dTMS) is one type of neuromodulation technique, and utilizing an H7 coil design can reach the dACC. Monitoring periodically throughout the first 6 months following treatment is crucial, given relapse within the first 6 months of treatment is robustly related to poor psychosocial functioning over the ensuing 1-3 years. The ultimate goal of this proposal is to provide treatment that more effectively promotes sustained abstinence in the Veteran with AUD, as extended abstinence is robustly associated with optimum biomedical, neuropsychological, psychiatric, and psychosocial recovery and functioning.

ELIGIBILITY:
Inclusion Criteria:

* The study will be open to male and females, regardless of race and ethnic origin, 21-70 years of age, who are in active treatment for an AUD at the VAPAHCS, Foundations of Recovery.
* Participants must meet Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria for AUD, and alcohol is self-identified as the primary substance of misuse.
* Able to read, verbalize understanding, and voluntarily sign the Informed Consent Form prior to participation in study procedures in English.
* Participants will be accepted if taking medications specifically for the treatment of major depressive disorders, cigarette smoking, or for other psychiatric conditions as long as the medications are not documented to lower seizure threshold - it would be clinically contraindicated to require participants to discontinue such medications for research. rTMS is safely administered to individuals who are taking psychotropic medications that do not lower seizure threshold.
* Participants will be abstinent from alcohol and non-prescribed substances for at least 7 consecutive days prior to rTMS to ensure no participant is experiencing active acute withdrawal.

Exclusion Criteria:

Psychiatric:

* Current diagnosis of Schizophrenia Spectrum Disorders and Bipolar Disorders;
* Current moderate-severe substance use disorder other than alcohol, tobacco, or marijuana, based on DSM-5 diagnostic criteria;
* Active current suicidal intent or plan (patients with a previous clinical flag for risk for suicide will be required to have an established safety plan involving their primary psychiatrist and the treatment team before entering the clinical trial, any form of previous rTMS or electroconvulsive treatment)

Biomedical:

Including, but not limited to:

* Uncontrolled thyroid disease,
* Unstable congestive heart failure,
* Angina
* Other severe cardiac illness as defined by treatment regimen changes in the prior 3 months
* Cerebrovascular accident, cancer if < 1 year since end of treatment;
* Unstable diabetes
* COPD requiring oxygen supplementation
* Alzheimer's disease
* Parkinson's disease
* Any biomedical implants with ferromagnetic content, neurostimulation devices, cardiac pacemakers or any magnetic resonance contraindications;
* Traumatic brain injury with self-reported or observed loss of consciousness > 30 minutes, any primary or traumatically induced seizure disorder, and alcohol-related seizure(s) in the past 30 days.

General:

* Lack of fluency in English;
* Wechsler Adult Reading Test below the 7th percentile (i.e., moderate or greater impairment in estimated general intelligence);
* Females who are pregnant or actively attempting pregnancy;
* Conservative exclusion for magnetic resonance research, current use of any medication or substance that is documented to lower seizure threshold or has been identified as a contraindication for rTMS treatment.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Padula, PhD, Principal Investigator — Stanford University; Michelle Madore, PhD, Principal Investigator — Stanford University; Timothy Durazzo, PhD, Principal Investigator — Stanford University
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Any data, specimens, forms, reports, and other records that leave the site will be identified only by a participant ID number to maintain confidentiality. The ID Number will have no relationship to any aspect of identifiable private information. Therefore, the data associated with each participant will be completely de-identified and there will be no mechanism by which users can re-identify participant data (e.g., name, address) with the subject code.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Three to twelve months after publication.
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Background] Koob GF, Volkow ND. Neurocircuitry of addiction. Neuropsychopharmacology. 2010 Jan;35(1):217-38. doi: 10.1038/npp.2009.110. PMID 19710631
- [Background] Peters SK, Dunlop K, Downar J. Cortico-Striatal-Thalamic Loop Circuits of the Salience Network: A Central Pathway in Psychiatric Disease and Treatment. Front Syst Neurosci. 2016 Dec 27;10:104. doi: 10.3389/fnsys.2016.00104. eCollection 2016. PMID 28082874
- [Background] Harel M, Perini I, Kampe R, Alyagon U, Shalev H, Besser I, Sommer WH, Heilig M, Zangen A. Repetitive Transcranial Magnetic Stimulation in Alcohol Dependence: A Randomized, Double-Blind, Sham-Controlled Proof-of-Concept Trial Targeting the Medial Prefrontal and Anterior Cingulate Cortices. Biol Psychiatry. 2022 Jun 15;91(12):1061-1069. doi: 10.1016/j.biopsych.2021.11.020. Epub 2021 Dec 6. PMID 35067356

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active dTMS
Started | 8
Received TMS Treatment | 6
Completed | 4
Not Completed | 4
Not completed — Withdrawal by Subject | 3
Not completed — Unable to complete preassessment MRI | 1

BASELINE CHARACTERISTICS:
Population: Participants who received TMS.
Arm/Group | Active dTMS
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Relapse to Alcohol 6 Months After Treatment
Description: Six months after completing the intervention, participants will be contacted to determine self-reported relapse status. To determine relapse status, participants complete brief standardized measures of alcohol and substance use, Alcohol Timeline Followback (TLFB) and the Brief Addiction Monitor (BAM) questionnaire.
Time Frame: 6 months
Population: Participants who completed at least half of the treatment sessions.
Measure: Count of Participants; unit: Participants
Arm/Group | Active dTMS
Number analyzed (Participants) | 5
Participants | 3

2. Primary Outcome: Percentage of Days Abstinent
Description: Abstinence defined as no drinks consumed.
Time Frame: 6 months
Population: Participants who completed at least half of the treatment sessions.
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Active dTMS
Number analyzed (Participants) | 5
percentage of days | 85.1 (32.06)

3. Primary Outcome: Percentage of Days of Heavy Drinking
Description: Heavy drinking is defined as consuming (in a 24 hour period) 3 or more drinks for women, or 4 or more drinks for men.
Time Frame: 6 months
Population: Participants who completed at least half of the treatment sessions.
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Active dTMS
Number analyzed (Participants) | 5
percentage of days | 2.7 (5.37)

ADVERSE EVENTS:
Time Frame: 10 days (TMS treatment) plus 6 months (follow-up)
Arm/Group | Active dTMS
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2022-06-28): https://cdn.clinicaltrials.gov/large-docs/64/NCT04927364/Prot_002.pdf